CLINICAL TRIAL: NCT06616805
Title: Effect of Low Volume High Intensity Interval Versus Moderate Intensity Continuous Training on Microalbuminurea in Patients With Diabetic Nephropathy
Brief Title: Effect of High Intensity Interval Versus Moderate Intensity Continuous Training on Microalbuminurea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Mohamed Ali Hussein, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004815
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: patients will be randomly assigned into two groups group A and group B. group A will receive low-volume high intensity interval training and group B will receive moderate intensity continuous training.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: quadruple (participant, care provider, investigator, outcome assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-volume High Intensity Interval Training (Experimental): Group (A): low-volume High Intensity Interval Training Patients in this group will undergo a warm-up at low intensity for 10 minutes, and then they will perform a single bout protocol that consisted of 1×4 min at 80-90% HRmax. Finally, a 5-min cool-down period will be permitted. The speed and the inclination of the treadmill will be adjusted to ensure that all patients are exercising at the desired target heart rate monitored by Pulse Oximeter.
  Interventions: Device: treadmill
- Moderate Intensity Continuous Training (Experimental): Group (B): Moderate Intensity Continuous Training Each session will start with a 10-minute warm-up at low intensity. Then they will walk on a treadmill for 30 min at moderate intensity corresponding to 65-75% of HR-max. Finally, a 5-min cool-down period will be permitted
  Interventions: Device: treadmill

INTERVENTIONS:
Device: treadmill — Treadmill JAGUAR treadmill:( T900, China) motorized treadmill model (T900) motor power (6.OHP) input voltage (AC220-240 V, 50Hz) speed range (1-20KM/H), inclination range (1-15%) was used for exercise treatment

SUMMARY:
purpose: to investigate the effect of low-volume high-intensity interval training and moderate- intensity continuous training on microalbuminuria in patients with diabetic nephropathy. methods: forty patients with microalbuminurea will be recruited and randomly assigned to two groups, group A and group B. patients in group A will receive low-volume HIIT and patients in group B will receive MICT. All patients will be evaluated pre and post treatment for laboratory investigation for ( HBa1c, ACR),and blood pressure.

DETAILED DESCRIPTION:
1. procedures for evaluation: the practical part of the study will be undertaken in 12 weeks(3 sessions a week).measurement will be taken before the start of treatment program then after the end of 12 weeks treatment program in the following manner:

   1. Anthropometric measures: body mass index (BMI) in kg/m2, waist circumference.
   2. Blood pressure measurement: Systolic and diastolic blood pressure.
   3. Biochemical (Lab) analysis:HbA1c, Urinary albumin test (Albumin/Creatinine ratio).
   4. Treadmill Graded exercise test:(Modified Bruce protocol) It will be used before starting of exercise sessions to determine maximum heart rate reached during this test and to predict individualized training target heart rate and training intensity for each patient before training.
2. Treatment procedures: All subjects in the exercise groups A&B will perform the exercise interventions using a treadmill 3 sessions per week for 12 weeks. In the early beginning, patients in all groups will receive an educational session about dietary guidelines for type 2 diabetes.

Group (A): low-volume High Intensity Interval Training Patients in this group will undergo a warm-up at low intensity for 10 minutes, and then they will perform a single bout protocol that consisted of 1×4 min at 80-90% HRmax. Finally, a 5-min cool-down period will be permitted. The speed and the inclination of the treadmill will be adjusted to ensure that all patients are exercising at the desired target heart rate monitored by Pulse Oximeter.

Group (B): Moderate Intensity Continuous Training Each session will start with a 10-minute warm-up at low intensity. Then they will walk on a treadmill for 30 min at moderate intensity corresponding to 65-75% of HR-max. Finally, a 5-min cool-down period will be permitted.

ELIGIBILITY:
Inclusion Criteria:

- 1. Type II diabetes mellitus 2. Age between 40 to 55 years old. 3. Blood pressure less than or equals 160/100 mmHg. 4. Patients receiving oral hypoglycemic. 5. Increased urinary albumin excretion (UAE)in the absence of other renal diseases.

6. Microalbuminuria (UAE >30µg /min and <299µg /min)

Exclusion Criteria:

* 1. Patients with Cardiac diseases. 2. Patients with chest diseases (Bronchial asthma and chronic obstructive pulmonary disease).

  3. Patients with severe self-limiting illness(cancer). 4. Musculoskeletal or neurological limitations to physical exercise. 5. Patients using insulin therapy. 6. Patients with poorly controlled DM (HbA1c > 9%). 7. Systolic Blood pressure more than 160 mmHg. 8. Morbid obesity. 9. Severe neuropathy. 10. PAD (claudication). 11. Retinopathy (moderate /advanced).

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
albumin/creatinine ratio | change in 12 weeks
  Random urine samples will be collected from patients before and after the end of treatment sessions for measuring al/Cr ratio
Glycated hemoglobin | change in 12 weeks
  blood samples will be collected from patients before and after the end of treatment sessions for measuring HBA1C

SECONDARY OUTCOMES:
blood pressure | change in 12 weeks
  Mercury sphygmomanometer (ALPK2, Japan) was used to measure systolic and diastolic blood pressure before exercise and after the end of treatment sessions

CONTACTS AND LOCATIONS:
Overall Officials: Heba Ali Abd El Ghafar, A.professor, Study Director — Cairo University
Locations (1):
- faculty of physical therapy, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No